CLINICAL TRIAL: NCT06846346
Title: Phase II Study Evaluating Ivonescimab in Combination With Chemotherapy for First- and Second-line Treatment of Advanced or Metastatic Gastric and Gastroesophageal Adenocarcinoma Patients
Brief Title: Testing Ivonescimab in Combination With Chemotherapy in Advanced or Metastatic Gastric/Gastroesophageal Adenocarcinoma
Acronym: GRACIE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2411; 2025-520694-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Esophageal Adenocarcinoma; Advanced Esophageal Adenocarcinoma; Metastatic Gastric Adenocarcinoma; Advanced Gastric Adenocarcinoma
Keywords: Ivonescimab; Esophageal; Gastric; Adenocarcinoma; Cancer; Metastatic; Advanced; FOLFOX; Irinotecan; Paclitaxel
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Adenocarcinoma; Neoplasms; Neoplasm Metastasis | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st line (Experimental): FOLFOX combined with Ivonescimab
  Interventions: Drug: Ivonescimab; Drug: FOLFOX regimen
- 2nd line (Experimental): Paclitaxel or Irinotecan (at investigator discretion) combined with ivonescimab
  Interventions: Drug: Ivonescimab; Drug: Irinotecan; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ivonescimab — Ivonescimab 20 mg/kg by intravenous (IV) infusion once every 2 weeks until disease progression.
  Other Names: AK112
Drug: FOLFOX regimen — Oxaliplatin 85 mg/m2 IV, folinic acid 400 mg/m2 IV (or L-folinic acid 200 mg/m²), and fluorouracil (5-FU) 400 mg/m² IV bolus; followed by 5 FU 2400 mg/m2 as a 46 hour continuous IV infusion, every two weeks for 8 cycles followed by 5FU as maintenance therapy until disease progression.
  Other Names: Oxaliplatin, folinic acid and 5-FU
  Arms: 1st line
Drug: Irinotecan — 180 mg/ m2 IV over 90 min infusion every two weeks for a minimum of 4 cycles
  Other Names: Campto
  Arms: 2nd line
Drug: Paclitaxel — 80 mg/m2 IV at D1, D8 and D15, every four weeks (D1=D28)
  Other Names: Taxol
  Arms: 2nd line

SUMMARY:
The goal of this clinical trial is to evaluate the addition of ivonescimab to standard chemotherapy in patients with advanced or metastatic gastric and gastroesophageal adenocarcinoma. The main question it aims to answer is : Does the addition of ivonescimab increase the response to treatment ? Participants will visit the clinic every 2 weeks for checkups, treatment administration and tests for collection of adverse events.

DETAILED DESCRIPTION:
Phase 2, multicenter, two-cohort, non-randomized, open-label trial to evaluate the efficacy of ivonescimab in combination with chemotherapy in patients with advanced or metastatic gastric and esophageal adenocarcinoma, with and without actionable biomarker (HER2/PD-L1/claudin18.2).

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form prior to any trial specific procedures. Note: If the patient is physically unable to provide their written consent, a trusted person of their choice, independent of the Investigator or the Sponsor, can confirm the patients consent in writing.
2. Histologically or cytologically proven gastric cancer (GC) or esophagogastric junction cancer adenocarcinoma (EGJC)
3. Metastatic or locally advanced non resectable (stage IV) disease.
4. Presence of at least one measurable lesion as assessed by the investigator according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Age ≥18 years.
7. For patients without actionable biomarker (HER2 and Claudin 18.2-negative) except for PD-L1, no prior treatment for advanced disease (cohort 1). For patients with at least one of the following actionable biomarker (PD-L1 CPS≥1, and/or HER2-positive, and/or Claudin 18.2-positive), who had received only one prior line of treatment for advanced disease (cohort 2).
8. Adequate hematological function: absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, platelet count ≥100 × 10⁹/L, and hemoglobin ≥9 g/dL. Note: Blood transfusion or growth factor therapy should not be performed within 7 days prior to the screening hematology analysis.
9. Adequate renal function: estimated creatinine clearance ≥50 mL/min according to the Cockcroft-Gault formula, or estimated glomerular filtration rate (eGFR) value ≥50 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, and urine protein < 2+ or 24-hour urine protein quantification < 1.0 g.
10. Adequate liver function: total bilirubin level ≤1.5 × the upper limit of normal (ULN) range (≤3 x ULN for patients with liver metastases or confirmed/suspected Gilbert syndrome), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 × ULN (AST and ALT ≤5 x ULN when documented liver metastasis).
11. Coagulation: prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy).This applies only to patients who are not on therapeutic anti-coagulation. Patients receiving therapeutic anti-coagulation should be on a stable dose.
12. Women of childbearing potential (WOCBP) having sex with an unsterilized male partner and unsterilized males having sex with a female partner of childbearing potential, must agree to use an effective method of contraception for the duration of trial participation and as required after completing study treatment (120 days after the last dose of ivonescimab). Men must also agree to not donate sperm and women must agree to not donate oocytes during the specified period.
13. WOCBP must have a negative serum pregnancy test performed within 3 days before inclusion and a negative urine pregnancy test on the day of first dose, prior to treatment administration.
14. Willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests, and other study procedures
15. Affiliation to the Social Security System (or equivalent)

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from gastroesophageal cancer within 2 years prior to study inclusion, except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (lamina propria invasion)].
2. Patients with high microsatellite instability (MSI-H) or mismatched repair disease (dMMR) tumor.
3. Enteral intake < 1500 kcal /d and or a weight loss > 15% of total body weight within the 6 months
4. Toxicities from previous treatment not resolved to grade ≤ 1 (according to the version 5.0 of the National Cancer Institute - Common terminology criteria for adverse events [NCI-CTCAE v5.0]) before treatment start with the exception of alopecia.
5. Major surgical procedures or serious trauma within 4 weeks prior to treatment start, or plans for major surgery within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to treatment start.
6. History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to inclusion, including but not limited to:

   1. Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots), Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.
   2. Nasal bleeding /epistaxis (bloody nasal discharge is allowed),
   3. Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to treatment start is not allowed. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution.
7. Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy.
8. History of major diseases before inclusion, specifically:

   1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association classification ≥ grade 2) or unstable vascular disease (eg, aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 12 months prior to inclusion, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia),
   2. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before inclusion,
   3. History of any grade arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in NCI-CTCAE v5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to inclusion,
   4. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before inclusion,
   5. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to inclusion.
9. Imaging during the screening period shows that the patient has:

   1. Radiologically documented evidence of major blood vessel invasion or encasement by cancer,
   2. Radiographic evidence of intra-tumor cavitation.
   3. Evidence of higher bleeding risk on prostheses
10. Any immunosuppressive therapy during more than 7 days (i.e. corticosteroids >10mg or equivalent dose) within 14 days before the planned start of study therapy. Physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is not considered as a form of systemic treatment.
11. Active autoimmune disease that has required a systemic treatment in past 2 years (i.e. corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin) is allowed active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study,
    2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study,
    3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    I. Rash must cover < 10% of body surface area, II. Disease is well controlled at baseline and requires only low-potency topical corticosteroids, III. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
12. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
13. Known history of, or any evidence of, interstitial lung disease.
14. Patient with non-controlled human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) infection (patient with undetectable viral load (HIV RNA PCR) and CD4 above 350 either spontaneously or on stable anti-viral regimen).
15. Chronic hepatitis B or C infection (if hepatitis status cannot be obtained from medical records, re-testing is required)
16. In case of planned treatment with fluorouracil, proven complete deficiency of dihydropyrimidine dehydrogenase (DPD).
17. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
18. Pregnant or breast-feeding females.
19. Participation in another therapeutic trial within the 30 days prior to entering the study. Participation in an observational trial would be acceptable.
20. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.
21. Individuals deprived of liberty or placed under protective custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate assessed by central review | Time from randomization to disease progression, up to 3 years
  The objective response rate is defined as the percentage of patients with a complete response (CR) or a partial response (PR) for a given treatment

SECONDARY OUTCOMES:
Objective Response Rate assessed by the investigator | Time from randomization to disease progression, up to 3 years
  The objective response rate is defined as the percentage of patients with a complete response (CR) or a partial response (PR) for a given treatment
Duration of response | Time from randomization to disease progression or death, up to 3 years
  The time form first documented response (compared to baseline measurement taken at randomization) until the date of disease progression or death from any cause, whichever occurs first
Progression-free survival (PFS) | Time from randomization to disease progression or death, up to 3 years
  The progression-free survival is the lengh of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse
Overall Survival (OS) | From randomization to death from any cause, up to 3 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Time to patient performance status deterioration >2 | From randomization to PS deterioration >2, up to 3 years
  Time to performance status (PS) deterioration >2 is defined as the time between patient randomisation and the first date when PS>2.
  The Eastern Cooperative Oncology Group (ECOG) PS, a simple measure of functional status, determines ability of patient to tolerate therapies. It has scores ranging from 0 to 5 (0 = "fully active", 1 = "completely ambulatory", 2 = "<50% in bed during the day", 3 = ">50% in bed, but not bedbound", 4 = "bedbound", and 5 = "death").
Incidence of Treatment Adverse Events | Throughout study completion, up to 3 years
  The tolerance and safety will be evaluated by toxicity (acute [<1 months after the end of the trial treatment] and late [≥1 month after the end of the trial treatment), assessed using the Common terminology criteria for adverse events version 5.0 (CTCAE v5.0). CTCAE is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 2 months, 6 months, disease progression and first follow-up visit (up to 3 years).
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Oesophago-Gastric cancer (QLQ-OG25) | At baseline, 2 months, 6 months, disease progression and first follow-up visit (up to 3 years).
  This EORTC oesophago-gastric cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-OG25 contains 25 items organized into six scales: dysphagia (three items), eating restrictions (four items), reflux (two items), odynophagia (two items), pain and discomfort (two items) and anxiety (two items), and ten single items: eating in front of others, dry mouth, trouble with taste, body image, trouble swallowing saliva, choked when swallowing, trouble with coughing, trouble talking, weight loss and hair loss. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle DE LA FOUCHARDIERE, Principal Investigator — Institut Paoli-Calmettes; Judith RAIMBOURG, Principal Investigator — ICO - Site Renée Gauducheau
Locations (4):
- France (4):
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Jean Godinot, Reims
  - Institut de Cancerologie de l'Ouest - Site René Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.